CLINICAL TRIAL: NCT02411747
Title: Simulation-based Training for Flexible Cystoscopy - a Patient Transfer Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sarah Hjartbro Bube, Medical Doctor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H-4-2014-122
Record Dates: First submitted 2015-03-31; First posted 2015-04-08 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Education
Keywords: Medical; Urology; Randomized Controlled Trial; Endoscopy; Cystoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testing+endoscopic simulation training (Experimental): Endoscopic training in flexible cystoscopy by directed self-regulated training with knowledge of a test afterwards, max. time cap 1h45min. 15 minutes of testing with a expert in the procedure. Total max time: 2 hours.
  Interventions: Behavioral: Testing; Behavioral: Directed self-regulated simulation training
- Oral lecture+endoscopic simulation training (Active Comparator): Endoscopic training in flexible cystoscopy by directed self-regulated training, max. time cap 1h45min after a 15 minute oral theoretical lecture by a expert in the procedure. Total max. time: 2 hours.
  Interventions: Behavioral: Directed self-regulated simulation training

INTERVENTIONS:
Behavioral: Testing
  Arms: Testing+endoscopic simulation training
Behavioral: Directed self-regulated simulation training

SUMMARY:
Simulation training in surgical education in Urology specialist training in flexible cystoscopy has been demonstrated a valid and efficient learning instrument. The classical setup with a medical expert introducing the novices to the theoretical background and technics of the procedure is time-consuming and expensive. Directed self-regulated simulation training (DSR) is a validated method in simulation training. The power of testing in DSR and flexible cystoscopy is to our knowledge not known. We introduced a setup in which the novices started by training in a directed self-regulated simulation training environment and informed them that they would be tested by a medical expert afterwards. The intervention group novices were given only written theoretical information and anatomical pictures. The control group were first given a classical oral theoretical introduction by a medical expert and secondly did DSR training. We tested the outcome of the intervention by a validated rating scale for flexible cystoscopy. The novices in both the control and intervention group were tested on patients prescribed a flexible cystoscopy and evaluated by a specialist in Urology.

The main hypothesis was that testing in relation to DSR would result in higher scores on a validated scale when performing a flexible cystoscopy on a patient evaluated by a specialist in Urology compared to a group having a oral lecture before DSR.

ELIGIBILITY:
Inclusion Criteria:

* Senior medical students
* Novices in endoscopic procedures
* Written and oral consent

Exclusion Criteria:

* Performed a endoscopic procedure independently
* Lack of language skills
* Lack of written and oral consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah H. Bube, Cand.med., Principal Investigator — Rigshospitalet, Denmark

REFERENCES:
- [Background] Matsumoto ED, Hamstra SJ, Radomski SB, Cusimano MD. A novel approach to endourological training: training at the Surgical Skills Center. J Urol. 2001 Oct;166(4):1261-6. doi: 10.1016/s0022-5347(05)65749-7. PMID 11547054
- [Background] Schout BM, Ananias HJ, Bemelmans BL, d'Ancona FC, Muijtjens AM, Dolmans VE, Scherpbier AJ, Hendrikx AJ. Transfer of cysto-urethroscopy skills from a virtual-reality simulator to the operating room: a randomized controlled trial. BJU Int. 2010 Jul;106(2):226-31; discussion 231. doi: 10.1111/j.1464-410X.2009.09049.x. Epub 2009 Nov 12. PMID 19912184
- [Background] Kromann CB, Jensen ML, Ringsted C. The effect of testing on skills learning. Med Educ. 2009 Jan;43(1):21-7. doi: 10.1111/j.1365-2923.2008.03245.x. PMID 19140995
- [Background] Brydges R, Nair P, Ma I, Shanks D, Hatala R. Directed self-regulated learning versus instructor-regulated learning in simulation training. Med Educ. 2012 Jul;46(7):648-56. doi: 10.1111/j.1365-2923.2012.04268.x. PMID 22691145
- [Background] Persoon MC, Schout BM, Muijtjens AM, Hendrikx AJ, Witjes JA, Scherpbier AJ. The effect of a low-fidelity model on cystoscopic skill training: a single-blinded randomized controlled trial. Simul Healthc. 2010 Aug;5(4):213-8. doi: 10.1097/SIH.0b013e3181e1b73d. PMID 21330799
- [Derived] Bube S, Dagnaes-Hansen J, Mahmood O, Rohrsted M, Bjerrum F, Salling L, Hansen RB, Konge L. Simulation-based training for flexible cystoscopy - A randomized trial comparing two approaches. Heliyon. 2020 Jan 3;6(1):e03086. doi: 10.1016/j.heliyon.2019.e03086. eCollection 2020 Jan. PMID 31922043

RESULTS

PARTICIPANT FLOW:
Groups:
- Directed Self-regulated Simulation Training+Testing: Endoscopic training in flexible cystoscopy by directed self-regulated training with knowledge of a test afterwards, max. time cap 1h45min. 15 minutes of testing with an expert in the procedure. Total max time: 2 hours.
  Directed self-regulated simulation training Testing
- Oral Lecture+Simulation Training: Endoscopic training in flexible cystoscopy simulation training, max. time cap 1h45min after a 15 minute oral theoretical lecture by an expert in the procedure. Total max. time: 2 hours.
  Oral expert lecture Simulation training
Period: Overall Study
Arm/Group | Directed Self-regulated Simulation Training+Testing | Oral Lecture+Simulation Training
Started | 16 | 16
Simulation Training Completed | 16 | 16
Completed | 13 | 12
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Directed Self-regulated Simulation Training+Testing: Endoscopic training in flexible cystoscopy by directed self-regulated training with knowledge of a test afterwards, max. time cap 1h45min. 15 minutes of testing with a expert in the procedure. Total max time: 2 hours.
  Directed self-regulated simulation training Testing
- Oral Lecture+Simulation Training: Endoscopic training in flexible cystoscopy by simulation training, max. time cap 1h45min after a 15 minute oral theoretical lecture by a expert in the procedure. Total max. time: 2 hours.
  Oral expert lecture Simulation training
- Total: Total of all reporting groups
Arm/Group | Directed Self-regulated Simulation Training+Testing | Oral Lecture+Simulation Training | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 26 [25 to 30] | 26 [24 to 31] | 26 [24 to 31]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 3 | 5 | 8
Future interest for surgical specility [Number; unit: participants]
  Surgical | 10 | 9 | 19
  Not surgical/not desided | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Global Rating Scale
Description: The subjects perform a flexible cystoscopy on two different patients and each cystoscopy are being scored by a specialist in Urology (the same in the entire study) using a validated scoring system for flexible cystoscopy, the Global Rating Scale. A previously validated assessment tool, Global Rating Scale (GRS) was used to assess the cystoscopy procedures. GRS is composed of five different parameters: respect for tissue, time and motion, handling of endoscope, flow of procedure, forward planning, and knowledge of procedure. Each parameter is assessed on a five point Likert scale with a minimum of one to maximum of five, giving the total GRS score a range of five to 25. At our institution we have defined a GRS score of three in each parameter (minimum total GRS of 15) as a minimum passing standard.
Time Frame: Two to four weeks after day of simulation training
Population: Two cystoscopies performed on patients by each participant
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Number cystoscopies
Arm/Group | Directed Self-regulated Simulation Training+Testing | Oral Lecture+Simulation Training
Number analyzed (Participants) | 13 | 12
Number analyzed (Number cystoscopies) | 26 | 24
units on a scale | 13.6 (4.2) | 13.4 (3.4)
Statistical Analysis 1: Comparison: Directed Self-regulated Simulation Training+Testing vs Oral Lecture+Simulation Training; Independent samples t-test; Test type: Non-Inferiority or Equivalence — Beta: 0.8, p significant if p > 0.005; p = 0.34, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Directed Self-regulated Simulation Training+Testing | Oral Lecture+Simulation Training
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes